CLINICAL TRIAL: NCT07267013
Title: Clindamycin as an Alternative to Vancomycin in Patients Undergoing Aortic Cardiac Surgery With Extracorporeal Circulation (ECC): a Prospective Single-center Pharmacokinetic Study
Brief Title: Clindamycin as an Alternative to Vancomycin in Patients Undergoing Aortic Cardiac Surgery With Extracorporeal Circulation (ECC)
Acronym: CLINDAPASS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RC24_0549; 2025-521555-23-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Aortic Surgery; Extracorporeal Circulation
Keywords: clindamycin; extracorporeal circulation (EEC); antibiotics
MeSH Terms: interventions — Clindamycin

STUDY DESIGN:
Intervention Model Description: Phase 2 interventional study, single-center, prospective and uncontrolled study conducted at Nantes University Hospital in the CTCV (Thoracic and Cardiovascular Surgery) anesthesia and intensive care unit.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clindamycin (Experimental)
  Interventions: Drug: Clindamycin

INTERVENTIONS:
Drug: Clindamycin — Clindamycin used in the study corresponds to commercial forms of injectable clindamycin : KBI 600 mg/4 mL injectable solution, ampoule.
  * 1 ampoule contains 600 mg Clindamycin phosphate (expressed as Clindamycin base).
  * Excipients: edetate disodium, benzyl alcohol, sodium hydroxide, water for injection.
  * Dosage form: injectable solution 10minutes after injecting the first bolus of cefuroxime, clindamycin is reconstituted in 50 mL of 0.9% NaCl, then 900 mg of clindamycin is administered as a slow IV over 30 minutes. At H+4 from the end of the clindamycin injection, if skin closure is not effective, clindamycin at a dose of 600 mg in 50 mL 0.9% NaCl is re-injected over 20 minutes.

SUMMARY:
Antibiotic prophylaxis is essential for all types of cardiac surgery under Extracorporeal Circulation (ECC), in order to reduce the incidence of surgical site infection (SSI). However, many patients are allergic to beta-lactam antibiotics. All the more, vancomycin antibiotic recommended as replacement is not without adverse effects and frequently administered in an inappropriate manner in terms of pre-intervention timing, linked to its complex use on peripheral venous lines complicated by venotoxicity. Non-compliance with the correct use of antibiotic prophylaxis in surgery is responsible for nosocomial infections, which have an impact on both the patient and the healthcare establishment in terms of costs, particularly in cardiac surgery.

Drug pharmacokinetics are more complex under bypass surgery (high volume of distribution), and studies are needed to determine the correct administration and diffusion of drugs.

In this respect, clindamycin is an antibiotic already used in antibiotic prophylaxis for other surgeries (thoracic, orthopedic...) in cases of allergy to beta-lactam antibiotics, but to date there are no studies examining the pharmacokinetics of this molecule in the context of cardiac surgery under ECC.

The aim of this protocol is to demonstrate the feasibility of using clindamycin in patients undergoing ECC surgery, by verifying that the plasma concentration of clindamycin exceeds the minimum inhibition concentration (MIC) of the main bacteria involved in mediastinitis throughout the surgical procedure.

DETAILED DESCRIPTION:
ECC is indispensable for cardiac surgery, but this assistance modifies the pharmacological properties of drugs, with a particular increase in the volume of distribution of antibiotics such as clindamycin. All these factors lead to an increase in the dosage of certain drugs and more frequent injections.

Robust data on percutaneous clindamycin treatment would therefore enable to improve the management of this type of patient, with real impact.

There are currently no pharmacological studies justifying the use of clindamycin to combat nosocomial infections in cardiac surgery, despite the fact that its anti-bacterial spectrum is identical to that of the antibiotics currently used in patients (methicillin-sensitive Staphylococcus aureus (MSSA)).

Clindamycin is simpler to use and does not induce venotoxicity. The fact that the patient is undergoing bypass surgery means that pharmacokinetic studies can be carried out with several blood samples taken from the arterial pressure catheter routinely inserted in all surgical patients, in order to limit the volume of blood taken and avoid any discomfort for the patient. This would make it possible to check the plasma stability of this antibiotic over several periods, with reinjections if necessary (if surgery > 4h).

The hypotheses are that clindamycin (i) is simple to use, (ii) has correct and stable diffusion kinetics in patients undergoing scheduled cardiac surgery with ECC (iii) is well tolerated by patients (iv) has an estimated free plasma concentration above the epidemiological threshold Minimal Inhibition Concentration (MIC) of Staphylococcus aureus and therefore provides sufficient protection against SSI.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 18 years of age,
* Cardiac surgery under ECC
* Surgery scheduled in the morning (added to the schedule at least 24 hours before the operation and starting at 8 a.m. in order to send blood tests during working hours).
* Written, informed consent from the patient before the start of the protocol.
* The patient must understand spoken and written French
* Negative pregnancy test and effective contraception (according to CTFG recommendations) during treatment for women of childbearing age
* Men of reproductive age using effective contraception (according to CTFG recommendations) during treatment
* Social security affiliation
* Patient able to understand the objectives of the study and comply with the requirements of the protocol

Exclusion Criteria:

* Known hypersensitivity/allergy to clindamycin, lincomycin, and any other excipient listed in the SmPC
* Known hypersensitivity/allergy to penicillins/drugs of the beta-lactam family
* Patient on antibiotics other than cefazolin prior to surgery
* Patient already on clindamycin at inclusion,
* BMI>35
* Aortic arch surgery
* Coronary artery bypass graft surgery
* Surgery for suspected endocarditis
* Patients with chronic renal failure with creatinine clearance < 60 mL/min and/or undergoing chronic dialysis
* Patients with hepatic insufficiency (prothrombin rate<50% excluding anticoagulant therapy) or Child B and C cirrhosis
* Immunosuppressed patients receiving triple antiviral therapy
* Pregnant or breast-feeding women
* Women or men of childbearing age without effective contraception
* Serious, uncontrolled concomitant bacterial infections (e.g. septic shock)
* Patients deprived of their liberty by judicial or administrative decision (guardianship, curatorship, safeguard of justice)
* Patient not registered with social security
* Participation in any other therapeutic study with an exclusion period still in effect at the time of inclusion, or planned participation in another therapeutic study while taking clindamycin
* Contraindications to cefazolin or any of the ancillary treatments
* Mental state rendering the patient incapable of understanding the entire study
* Patient being the investigator or any other member of the research team or being a relative of the investigator directly involved in the trial, including assistant physicians, pharmacists, nurses, and study coordinators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-03-30 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Plasma clindamycin concentrations | H0 (at incision), then every hour, and at the end of surgery (defined as sternal closure)
  To demonstrate the feasibility of using clindamycin in patients undergoing ECC and to assure that plasma clindamycin concentrations remain above the minimum inhibition concentration (MIC) of the main bacteria involved in mediastinitis, estimated free plasma clindamycin concentration will be verify throughout surgery. The free plasma concentration of clindamycin is estimated by measuring the total plasma concentration of clindamycin, based on a bound fraction of 80 to 94%.The epidemiological threshold MIC for S. aureus (ECOFF = 0.25 mg/L for clindamycin) was chosen for comparison with clindamycin concentrations, given that this bacterium is the main one implicated in mediastinitis.

SECONDARY OUTCOMES:
Determine the pharmacokinetic parameters of clindamycin under ECC | At H0 (at incision), then every hour, and at the end of surgery (defined as sternal closure)
  Volume of distribution, clearance, elimination half-life, quantity of intra-operative vascular filling (in ml) including blood transfusions: number and type of intra-operative LBS (labile blood products)
Determine the factors of variability in clindamycin pharmacokinetics for patients under ECC surgery | Post-ECC at H+6 and H+24
  Collection of weight, height (calculation of BMI), collection of usual post-CEC biological data (creatinemia with calculation of GFR, ASAT/ALAT, total and conjugated bilirubinemia, PAL, γ-GT, protidemia with addition of α-1 acid glycoprotein at induction), qualitative record of CYP3A4/5 inducer/inhibitor drugs, CEC modalities (duration, type and quantity of priming solution, type of cardioplegia, body temperature), blood transfusion and volume reprocessed by Cell-Saver©.
Determining the diffusion of clindamycin in pericardial fatty tissue | At the start of the operation (sternotomy) and when the pericardium is closed
  Tissue determination of clindamycin in pericardial fat and correlation with plasma levels (biocollection, ancillary study
Description of adverse events according to NCI CTCAE V5 criteria | From first injection of clindamycin to end of hospitalization
  Recording of AEs and SAEs, collection of all clinical signs indicative of anaphylaxis on medical examination
Adherence to Good Clinical Practice clindamycin injection protocol | From first injection of clindamycin to the end of surgery (defined as sternal closure)
  Recording of clindamycin injection duration, time of reinjections and duration of reinjections, calculation of delta between time of end of clindamycin injection and start of surgical incision
Rate of post-operative mediastinitis (up to 3 months post-operatively) | From inclusion to 3 months post-operatively (M3)
  Rate of post-operative mediastinitis defined as a post-operative nosocomial cardiac surgery infection at the surgical site (mediastinum) requiring repeat surgery (drainage lavage) and prolonged antibiotic therapy. Collection of data from the patient's file, as the patient was systematically referred to the Nantes University Hospital. Collection of bacterial ecology
Post-op morbidity and mortality | At 3 months (M3) post-operative (follow-up)
  Mortality at 3 months (telephone call)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nantes, Nantes, France, France

IPD SHARING:
Plan to Share IPD: Undecided